CLINICAL TRIAL: NCT05110846
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multiple-Center Study to Evaluate the Efficacy, Safety, and Tolerability of CT-868 Administered for 26 Weeks to Overweight and Obese Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of CT-868 in Overweight and Obese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carmot Therapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-868-002; BP45664 (Other: Roche Protocol Number)
Record Dates: First submitted 2021-11-04; First posted 2021-11-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obesity; Overweight; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants in the placebo arm received volume- and regimen-matched placebo.
  Interventions: Drug: Placebo
- CT-868 1.75 mg (Experimental): Participants in the CT-868 1.75 mg arm received 1.0 mg/day for 2 weeks followed by 1.75 mg/day for the remaining treatment period.
  Interventions: Drug: CT-868
- CT-868 4.0 mg (Experimental): Participants in the CT-868 4.0 mg arm escalated through 1.0 mg/day for 2 weeks, 1.75 mg/day for 2 weeks, 2.5 mg/day for 4 weeks, 3.25 mg/day for 4 weeks, to 4.0 mg/day for the remaining 14 weeks.
  Interventions: Drug: CT-868

INTERVENTIONS:
Drug: Placebo — Participants self-injected once-daily subcutaneous volume- and regimen-matched placebo for 26 weeks.
  Arms: Placebo
Drug: CT-868 — Participants self-injected once-daily subcutaneous CT-868 for 26 weeks according to the randomized dose and regimen.
  Arms: CT-868 1.75 mg; CT-868 4.0 mg

SUMMARY:
A study to assess the effect of CT-868 in lowering glycated hemoglobin A1c (HbA1c) in overweight and obese participants with inadequately controlled Type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Males or Females with T2DM
* BMI of ≥27 kg/m2, inclusive
* 18-75 years old, inclusive
* Stable body weight for 3 months

Exclusion Criteria:

* Significant medical history
* Uncontrolled diabetes
* History of malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Glycated Hemoglobin A1c (HbA1c) at Week 26 | Baseline and Week 26

SECONDARY OUTCOMES:
Change from Baseline in HbA1c at Week 12 | Baseline and Week 12
Percentage of Participants Achieving HbA1c <5.7% at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percentage of Participants Achieving HbA1c ≤6.5% at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percentage of Participants Achieving HbA1c <7.0% at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percent Change from Baseline in Body Weight at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Absolute (kg) Change from Baseline in Body Weight at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percentage of Participants with ≥5% Body Weight Loss from Baseline at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percentage of Participants with ≥10% Body Weight Loss from Baseline at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percentage of Participants with ≥15% Body Weight Loss from Baseline at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percentage of Participants with ≥20% Body Weight Loss from Baseline at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Fasting Plasma Glucose at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Fasting Insulin at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Waist Circumference at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Hip Circumference at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Waist-to-Hip Ratio at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Waist-to-Height Ratio at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Body Mass Index (BMI) at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Total Cholesterol at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Triglycerides at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Low Density Lipoprotein (LDL) Cholesterol at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in High Density Lipoprotein (HDL) Cholesterol at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Very Low Density Lipoprotein (VLDL) Cholesterol at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Apolipoprotein B at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Change from Baseline in Quantitative Insulin Sensitivity Check Index (QUICKI) at Weeks 12 and 26 | Baseline and Weeks 12 and 26
Percentage of Participants with at Least One Treatment-Emergent Adverse Event | From first dose of study drug until 4 weeks after the last dose of study drug (30 weeks)
Percentage of Participants with at Least One Hypoglycemic Event | From first dose of study drug until 4 weeks after the last dose of study drug (30 weeks)
Percentage of Participants Testing Positive for Anti-Drug Antibodies to CT-868 at Baseline and Anytime Post-Baseline | Baseline and Post-Baseline (up to 30 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Carmot Therapeutics, Inc., a Member of the Roche Group
Locations (5):
- Mexico (5):
  - Carmot Clinical Center MX04, Guadalajara, Jalisco
  - Carmot Clinical Center MX01, Monterrey, Nuevo León
  - Carmot Clinical Center MX02, Monterrey, Nuevo León
  - Carmot Clinical Center MX05, Mérida, Yucatán
  - Carmot Clinical Center MX03, Mexico City

IPD SHARING:
Plan to Share IPD: No